CLINICAL TRIAL: NCT00833066
Title: Preliminary Assessment of the Clinical Tolerability, Safety and Immunogenicity of Three Different Doses of Grass Pollen-derived Peptides for Oral Use in Antigen-specific Immunotherapy of Seasonal Allergic Rhinoconjunctivitis
Brief Title: Safety Study of Grass Pollen-derived Peptides to Treat Seasonal Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioTech Tools S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTT-gpASIT003; EudraCT 2008-006369-10
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Seasonal Allergic Rhinoconjunctivitis
Keywords: hay fever; grass pollen allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- gpASIT 25 (Experimental)
  Interventions: Biological: gpASIT+TM
- gpASIT 100 (Experimental)
  Interventions: Biological: gpASIT+TM
- gpASIT 400 (Experimental)
  Interventions: Biological: gpASIT+TM

INTERVENTIONS:
Biological: gpASIT+TM — entero-coated capsules containing 25µg of gpASIT+TM
  Arms: gpASIT 25
Biological: Placebo — placebo entero-coated capsules
  Arms: Placebo
Biological: gpASIT+TM — entero-coated capsules containing 100µg of gpASIT+TM
  Arms: gpASIT 100
Biological: gpASIT+TM — entero-coated capsules containing 400µg of gpASIT+TM
  Arms: gpASIT 400

SUMMARY:
The purpose of this study is to determine whether the oral administration of grass pollen peptides is safe and effective in the treatment of allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent
* Age between 18 and 50 years
* The subjects are in good physical and mental health according to his/her medical history, vital signs, and clinical status
* Male or non pregnant, non-lactating female
* Female unable to bear children must have documentation of such in the CRF (i.e. tubule ligation, hysterectomy, or post menopausal (defined as a minimum of one year since the last menstrual period))
* Allergy:

A history of seasonal allergic rhinoconjunctivitis (SAR) during the grass pollen season during at least the two previous years A positive skin prick test (wheal diameter >= 3 mm) to grass-pollen mixture Specific IgE against grass pollen (RAST class 2 or IgE > 0.7 kU/l) Asymptomatic to perennial inhalant allergens.

Exclusion Criteria:

* Subjects with current or past immunotherapy (any time in the past)
* Subjects requiring controller medication against asthma (bronchodilator nebulised drugs or local or systemic corticosteroids)
* Documented evidence of acute or significant chronic sinusitis (as determined by individual investigator)
* Subjects with a history of hepatic or renal disease
* Subjects symptomatic to perennial inhalant allergens
* Subject with malignant disease, autoimmune disease
* Female subjects who are pregnant, lactating, or of child-bearing potential and not protected from pregnancy by a sufficiently reliable method (OCs, IUD)
* Any chronic disease, which may impair the subject's ability to participate in the trial (i.e. severe congestive heart failure, active gastric or duodenal ulcer, uncontrolled diabetes mellitus, etc…)
* Subjects requiring beta-blockers medication
* Chronic use of concomitant medications that would affect assessment of the effectiveness of the trial medication (e.g. tricyclic antidepressants)
* Subject with febrile illness (> 37.5°C, oral)
* A known positive serology for HIV-1/2, HBs antigen or anti-HCV antibodies
* The subject is immunocompromised by medication or illness, has received a vaccine, corticoids or immunosuppressive medications within 1 month before trial entry
* Receipt of blood or a blood derivative in the past 6 months preceding trial entry
* Regular consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 4 weeks preceding the trial
* Any consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 1 week preceding the trial
* Use of long-acting antihistamines
* Any condition which could be incompatible with protocol understanding and compliance
* Subjects who have forfeited their freedom by administrative or legal award or who are under guardianship
* Unreliable subjects including non-compliant subjects, subjects with known alcoholism or drug abuse or with a history of a serious psychiatric disorder as well as subjects unwilling to give informed consent or to abide by the requirements of the protocol
* Participation in another clinical trial and/or treatment with an experimental drug within 1 month of trial start
* A history of hypersensitivity to the excipients
* Rhinitis medicamentosa, non-specific rhinitis (to food dye, preservative agent…)
* Subjects without means of contacting the investigator rapidly in case of emergency, or not able to be contacted rapidly by the investigator
* Subjects who participated to trial BTT-gpASIT002

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evidence of allergic reaction | within the first 14 days (plus or minus 1 day)

SECONDARY OUTCOMES:
Immunological assessment | 9 months
Allergy symptom and medication scores | grass pollen season 2009

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - University Hospital Brugmann, Brussels
  - University Hospital Ghent, Ghent
  - University Hospital Gasthuisberg, Leuven
  - University Hospital Sart Tilman, Liège